CLINICAL TRIAL: NCT01771783
Title: Single-center, Randomized, Open-label, 3-way Crossover Study to Characterize the RAS-peptide-profile After Single and Repeated Oral Administration of Different RAS-inhibitors in Healthy Male Subjects
Brief Title: RAS-Peptide-Profile Study in Healthy Male Subjects
Acronym: RAS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: USBMH-001
Record Dates: First submitted 2013-01-16; First posted 2013-01-18 (Estimated); Last update posted 2013-05-13 (Estimated); Status verified 2013-05

CONDITIONS: RAS Peptide Profile in Healthy Volunteers
Keywords: RAS-Peptide Profile; Renin-Angiotensin-System; Angiotensin-Converting-Enzyme-Inhibitor; Angiotensin-Receptor-Antagonist; Renin-inhibitor
MeSH Terms: interventions — Angiotensin-Converting Enzyme Inhibitors; Angiotensin Receptor Antagonists; Renin Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- ACEI-ARB-RI (Experimental): angiotensin converting enzyme inhibitor (ACEI) angiotensin receptor antagonist (ARB) renin inhibitor (RI)
  Interventions: Drug: ACEI-ARB-RI; Drug: ARB-RI-ACEI; Drug: RI-ACEI-ARB
- ARB-RI-ACEI (Experimental): ARB-RI-ACEI
  Interventions: Drug: ACEI-ARB-RI; Drug: ARB-RI-ACEI; Drug: RI-ACEI-ARB
- RI-ACEI-ARB (Experimental): RI-ACEI-ARB
  Interventions: Drug: ACEI-ARB-RI; Drug: ARB-RI-ACEI; Drug: RI-ACEI-ARB

INTERVENTIONS:
Drug: ACEI-ARB-RI
  Other Names: angiotensin converting enzyme inhibitor (ACEI); angiotensin receptor antagonist (ARB); renin inhibitor (RI)
Drug: ARB-RI-ACEI
  Other Names: angiotensin converting enzyme inhibitor (ACEI); angiotensin receptor antagonist (ARB); renin inhibitor (RI)
Drug: RI-ACEI-ARB
  Other Names: angiotensin converting enzyme inhibitor (ACEI); angiotensin receptor antagonist (ARB); renin inhibitor (RI)

SUMMARY:
The primary objective is the characterization of the RAS peptide profiles after single and repeated oral administration of a renin inhibitor, an ACE inhibitor and an angiotensin receptor blocker in healthy volunteers.

Secondary objectives are the correlation of RAS peptide profiles with pharmacokinetic profiles of the different RAS inhibitors and with pharmacodynamic parameters such as blood pressure and heart rate. Output of the classic RAS system will be assessed using aldosterone concentrations. Fluid and sodium intake will be monitored using sodium concentration and total volume in 24h urine.

DETAILED DESCRIPTION:
The results of a pilot study have shown that single doses of different RAS inhibitors produce characteristic changes of the RAS peptide profiles. In a first step this finding needs to be verified in a larger number of healthy subjects. Since it is unknown, whether the changes that were observed within hours after a single inhibitor dose are stable over time, the profiles also need to be investigated under steady-state conditions of the different inhibitors. Comparison of RAS peptide profiles after single dose and under steady-state conditions will also allow to detect whether the peptide profiles are altered by compensatory mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Male aged between 18 and 45 years (inclusive) at screening.
* Body mass index (BMI) between 18 and 28 kg/m2 (inclusive) and body weight at least 50 kg at screening.
* Systolic blood pressure (SBP) 100-140 mmHg, diastolic blood pressure (DBP) 60-90 mmHg and heart rate (HR) 45-90 bpm (inclusive), measured on the leading arm*, after 5 min in the supine position at screening.
* Signed informed consent prior to any study-mandated procedure.
* No clinically significant findings on the physical examination at screening.
* 12-lead electrocardiogram (ECG) without clinically relevant abnormalities at screening.
* Hematology and clinical chemistry results not deviating from the normal range to a clinically relevant extent at screening.
* Ability to communicate well with the investigator and to understand and comply with the requirements of the study.

  * leading arm right = writing with right hand

Exclusion Criteria:

* Smoking > 5 cigarettes per day
* History or clinical evidence of alcoholism or drug abuse within the 3-year period prior to screening.
* Loss of ≥ 250 ml of blood within 3 months prior to screening.
* Treatment with an investigational drug within 30 days prior to screening.
* Previous treatment with any prescribed or over the counter medications (including herbal medicines such as St John's Wort) within 2 weeks prior to the intended start of study.
* Legal incapacity or limited legal capacity at screening.
* Positive results from urine drug screen at screening.
* History or clinical evidence of any disease and/or existence of any surgical or medical condition, which might interfere with the absorption, distribution, metabolism or excretion of the study drugs, or which might increase the risk for toxicity.
* Known hypersensitivity to any excipients of the drug formulations.
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2012-11; Primary Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
RAS-peptide profile | 0-192h

SECONDARY OUTCOMES:
Blood pressure and heart rate | 0-192 h
Aldosterone concentrations | 0-192 h

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Haschke, PD Dr. med., Principal Investigator — Clinical Pharmacology, University Hospital Basel
Locations (1):
- Department Clinical Pharmacology, University Hospital Basel, Basel, Switzerland